CLINICAL TRIAL: NCT05660967
Title: Efficacy and Safety of Epcoritamab Monotherapy and in Combination With Lenalidomide as First-line Therapy for Anthracycline-ineligible Diffuse Large B-Cell Lymphoma Patients, an Open-label, Randomized, Multicenter, Global Phase 2 Trial
Brief Title: Subcutaneous Epcoritamab With or Without Lenalidomide as First Line Therapy for Diffuse Large B-Cell Lymphoma
Acronym: EPCORE DLBCL-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-06; 2021-005744-29 (EudraCT Number); jRCT2021230015 (Registry Identifier: Japan Registry for Clinical Trials (jRCT)); 1006219 (Other: IRAS ID; UK Research Summaries Database); 2023-504832-16-00 (EU CTIS Number)
Expanded Access: NCT05733650 (Approved for marketing)
Record Dates: First submitted 2022-11-29; First posted 2022-12-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Double-hit lymphoma; Triple-hit lymphoma; Follicular grade 3B; T-cell/histiocyte rich LBCL; DuoBody®; Anti-CD3; Anti-CD20; Subcutaneous; Bispecific antibody; EPCORE
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epcoritamab monotherapy (Experimental)
  Interventions: Biological: Epcoritamab
- Epcoritamab in combination with lenalidomide (Experimental)
  Interventions: Biological: Epcoritamab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Epcoritamab — Epcoritamab will be administered by subcutaneous (SC) injections in 28-day cycles for up to 12 cycles.
  Other Names: GEN3013; DuoBody®-CD3×CD20; EPKINLY™
Drug: Lenalidomide — Lenalidomide will be administered orally (capsules; starting dose of 10 or 20 mg) once daily on Day 1 to Day 21 of each 28-day cycle for up to 12 cycles.
  Other Names: Revlimid®
  Arms: Epcoritamab in combination with lenalidomide

SUMMARY:
The purpose of the study is to examine efficacy and safety of epcoritamab with and without lenalidomide in newly diagnosed elderly patients with Diffuse Large B-Cell Lymphoma (DLBCL) who cannot tolerate anthracycline therapy. Epcoritamab (also known as EPKINLY™, GEN3013 and DuoBody®-CD3xCD20) is an antibody that has already been tested in several clinical studies. All patients will receive active treatment. There is an equal chance of receiving epcoritamab or epcoritamab plus lenalidomide.

DETAILED DESCRIPTION:
This is an open-label, multicenter, global phase-2 trial evaluating the efficacy and safety of epcoritamab monotherapy and epcoritamab plus lenalidomide in elderly patients who are deemed anthracycline ineligible.

The trial is designed in two stages:

* Stage 1 which includes a safety run-in phase in each arm
* Stage 2, an expansion of the selected treatment from Stage 1

ELIGIBILITY:
Inclusion Criteria:

* Must have newly diagnosed CD20+ large cell lymphoma.
* Is ineligible for anthracycline-based therapy/cytotoxic chemotherapy due to:

  * Being age ≥80 years; AND/OR
  * Being age ≥75 years and having important comorbid condition(s), which are likely to have a negative impact on tolerability of anthracycline-based therapy/cytotoxic chemotherapy.
* Have Immune Effector Cell-Associated Encephalopathy (ICE) score of at least 8 out of 10.
* Have Ann Arbor Stage II-IV disease.
* Have ECOG PS of 0, 1, or 2; (ECOG PS of 3 may be considered if impairment is attributed to current lymphoma/DLBCL and if pre-phase treatment during the screening phase results in an improvement of ECOG PS to ≤2 prior to enrollment).
* Have measurable disease as per Lugano criteria.
* Have acceptable organ function based on baseline bloodwork.
* Must have fresh (preferred) or archival biopsy material at screening.

Exclusion Criteria:

* Has known active, clinically significant bacterial, viral, fungal, mycobacterial, parasitic, or other infection at trial enrollment, including COVID-19 infection.
* Has severe cardiovascular disease (other than those eligibility criteria that preclude the subject from receiving anthracycline-based therapy/cytotoxic chemotherapy),
* Has been exposed to/received any of the following prior therapies, treatments, or procedures within the specified timeframes:

  * Major surgery within 4 weeks prior to the first dose of epcoritamab;
  * Non-investigational antineoplastic agents (except anti-CD20 monoclonal antibodies) or any investigational drug within 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of epcoritamab;
  * Autologous hematopoietic stem cell transplantation (HSCT), CAR-T, allogeneic stem cell transplantation, or solid organ transplantation;
  * Live, attenuated vaccines within 30 days prior to initiation of epcoritamab;
  * Investigational vaccines within 28 days before the planned first dose of epcoritamab (ie, experimental and/or non-authorized SARS-CoV-2 vaccinations and therapies are not allowed);
  * Invasive investigational medical device use within 28 days before the planned first dose of epcoritamab.
* Has primary central nervous system (CNS) tumor or known CNS involvement or intracranial involvement as confirmed by mandatory brain magnetic resonance imaging/computed tomography (MRI/CT) scan at screening and, if clinically indicated, by lumbar puncture.
* Has a seizure disorder requiring anti-epileptic therapy or experienced a seizure within 6 months of signing an informed consent form.
* Has known past or current malignancy other than inclusion diagnosis, with exceptions as stated in protocol.
* Has known or suspected allergies, hypersensitivity, or intolerance to either of the trial treatments or has known or suspected contraindication to the use of all locally available anti-cytokine therapies per local guidelines for management of cytokine release syndrome (CRS).
* Has active hepatitis B virus (HBV) (DNA polymerase chain reaction [PCR]-positive) or hepatitis C virus (HCV) (RNA PCR-positive) infection, current alcohol abuse, or cirrhosis.
* Has active cytomegalovirus (CMV) infection (DNA PCR-positive) requiring treatment.
* Has suspected active or inadequately treated latent tuberculosis.
* Has a known history of seropositivity for HIV. Note: HIV testing is required at screening only if required per local health authorities or institutional standards.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Percentage of participants achieving CR. Assessed by the Investigator per Lugano criteria

SECONDARY OUTCOMES:
Duration of response (DOR) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Defined as the time between date of first response to the date of first documented tumor progression or death (due to any cause) whichever occurs first
Duration of complete response (DOCR) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Defined as the time between the date of first CR to the date of the first documented tumor progression or death due to any cause, whichever comes first
Time to response (TTR) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 1 year
  Defined as the time from first dose to first documentation of objective tumor response (CR or PR)
Overall Response Rate (ORR) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Defined as the percentage of patients who achieve best overall response of complete response (CR) or partial response (PR) determined by Lugano criteria
Progression-free survival (PFS) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Defined as the time from first dose to date of PD or death (due to any cause) whichever occurs first
Time to next anti-lymphoma therapy (TTNT) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Defined as the time from first dose to administration of subsequent anti-lymphoma therapy
Rate of minimal residual disease (MRD) negativity | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 2 years
  Percentage of participants with at least 1 post-screening MRD negative result
Overall survival (OS) | From randomization (for patients enrolled in stage 1) or from first dose (for patients enrolled in stage 2) and up to 3 years
  Defined at the timeframe from first dose to death
Incidence and severity of adverse events (AEs) | From screening until end of the safety follow-up period (60 days after last dose)
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment
Incidence of clinically significant shifts in laboratory parameters | From screening until end of the safety follow-up period (60 days after last dose)
  Clinical laboratory parameters assessed: hematology, chemistry, coagulation, tumor lysis, cardiac enzymes, immunoglobulins, and urinalyses
Incidence of anti-drug antibodies (ADAs) to epcoritamab in plasma | From first dose until treatment discontinuation (assessed up to 12 months)
  To evaluate immunogenicity
Evaluate patient-reported outcomes (PROs) related to lymphoma symptoms | From cycle 1, day 1 until 90 days after last dose (each cycle is 28 days)
  Changes in lymphoma symptoms as measured by the Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym). Scale from 0-168 obtained by summing individual subscale scores. Higher scores for the scales indicate better quality of life
Assess pharmacokinetics (PK) of epcoritamab | From first dose and at multiple time points until treatment discontinuation (assessed up to 12 months)
  Total body clearance of drug from the plasma (CL)
Assess pharmacokinetics (PK) of epcoritamab | From first dose and at multiple time points until treatment discontinuation (assessed up to 12 months)
  Maximum observed concentration (Cmax)
Assess pharmacokinetics (PK) of epcoritamab | From first dose and at multiple time points until treatment discontinuation (assessed up to 12 months)
  Time to reach Cmax (Tmax)
Assess pharmacokinetics (PK) of epcoritamab | From first dose and at multiple time points until treatment discontinuation (assessed up to 12 months)
  Terminal Elimination Half-Life (t 1/2)

CONTACTS AND LOCATIONS:
Locations (74):
- UW Cancer Center at ProHealth Care, Waukesha, Wisconsin, United States
- Austria (3):
  - Kepler Universitätsklinikum, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - ZNA, Antwerp
  - UZ Brussels, Jette
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
  - Vitaz, Temse
  - AZ Turnhout - Campus Sint-Elisabeth, Turnhout
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (10):
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - Hôpital Henri Mondor, Créteil
  - Hopital Claude Huriez - CHRU Lille, Lille
  - Hopital de la Conception - APHM, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hôpital Saint-Antoine, Paris
  - Hôpital Saint-Louis, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - CHU Amiens - Hopital Sud, Salouël
  - CHU Tours - Hôpital Bretonneau, Tours
- Germany (4):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Aachen AOeR, Aachen
  - Vivantes Klinikum Neukoelln, Berlin
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (11):
  - Clinica di Ematologia AOU Ospedali Riuniti di Ancona, Ancona
  - IRCCS Centro di Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo
  - IRCCS Istituto Romagnolo Per Lo Studio Dei Tumori "Dino Amadori" - IRST, Meldola
  - IEO Istituto Europeo di Oncologia Parent, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - AUSL Piacenza Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda sanitaria integrata università di Trieste, Trieste
- Japan (9):
  - Kyushu University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Matsuyama Red Cross Hospital, Matsuyama
  - NHO Nagoya Medical Center, Nagoya
  - Kindai University Hospital, Ōsaka-sayama
  - Yamagata University Hospital, Yamagata
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Pratia MCM Krakow, Krakow
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - MICS Centrum Medyczne Torun, Torun
- South Korea (6):
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Jeonbuk National University Hospital, Jeonju
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (11):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Universitario Puerta del Mar, Seville
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (5):
  - Royal Marsden Hospital - Fulham, London
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton
  - Royal Cornwall Hospital NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: No